

# STATISTICAL ANALYSIS PLAN (SAP)

### **Non-Interventional Study Protocol**

A3921302

### **ESCALATE-RA**

A NON-INTERVENTIONAL STUDY OF CRITICAL FACTORS FOR ESCALATING DRUG TREATMENT IN PATIENTS TREATED WITH TOFACITINIB FOR MODERATE TO SEVERE ACTIVE RHEUMATOID ARTHRITIS

# Statistical Analysis Plan (SAP)

**Version**: Final v 2.0

Author: PPD

Date: 07-AUG-2023

### **TABLE OF CONTENTS**

| 1 | LIST OF ABBREVIATIONS6 |
|---|---|
| 2 | AMENDMENTS FROM PREVIOUS VERSION(S)7 |
| 3 | INTRODUCTION |
| | 3.1STUDY DESIGN93.2STUDY POPULATION113.2.1Treatment/cohort labels123.2.1.1Treatment Label for Secondary Analysis123.2.1.2Treatment Label for Secondary Analysis – Subgroup Sequence of Therapy123.3STUDY OBJECTIVES12 |
| 4 | INTERIM AND FINAL ANALYSES |
| | 4.1 Interim Analysis 13 4.2 Final Analysis 13 4.3 Pooled Analysis 13 |
| 5 | HYPOTHESES AND DECISION RULES |
| 6 | ANALYSIS SETS/ POPULATIONS |
| 7 | 6.1 ALL PATIENT SET 14 6.2 FULL ANALYSIS SET 14 6.3 SECONDARY FULL ANALYSIS SET 14 6.4 SAFETY ANALYSIS SET 14 6.5 PER PROTOCOL ANALYSIS SET 14 6.6 SUBGROUPS 15 ENDPOINTS AND COVARIATES 16 |
| 7 | |
| | 7.1 EFFICACY/ EFFECTIVENESS ENDPOINT(S) 16 7.1.1 Primary Endpoints 16 7.1.2 Secondary Endpoints 17 7.1.2.1 Time to first treatment escalation 17 7.1.2.2 Rate of LDA 18 7.1.2.2.1 SDAI LDA 18 7.1.2.2.2 CDAI LDA 18 7.1.2.2.3 DAS28-4 (ESR) LDA 19 7.1.2.3 Rate of Remission 19 7.1.2.3.1 ACR-EULAR Boolean remission criteria 20 7.1.2.3.2 SDAI Remission 20 7.1.2.3.3 CDAI Remission 20 |
| Fi | nal Version 07-AUG-2023 |

| | 7.1.2.3.4 DAS28-4 (ESR) Remission | . 21 |
|---|---|---|
| | 7.1.2.3.5 DAS28-4 (CRP) Remission | 21 |
| | 7.1.2.4 Change from Baseline in DAS28-4 (ESR) and DAS28-4 (CRP) | |
| | 7.1.2.5 Change from Baseline in Duration of Morning Stiffness | |
| | 7.1.2.6 Change from Baseline in FFbH | |
| | 7.1.2.7 Rate of Functional Remission (FFbH) | |
| | 7.1.2.7 Rate of Functional Refinssion (FF011) | |
| | 7.1.2.6 Change from Baseline in FACIT-Fatigue | |
| | $\mathcal{C}$ | |
| | 7.3 COVARIATES, FACTORS AND POTENTIAL CONFOUNDERS | |
| | 7.3.1 Factors of Interest for Primary Analysis | |
| | 7.3.2 factors of Interest for Sensitivity of the Primary Analysis | |
| | 7.3.3 Potential Confounders to be included in the Primary Analysis | . 21 |
| 8 | HANDLING OF MISSING VALUES | 29 |
| | 8.1 TIME TO EVENT (PRIMARY ANALYSIS, TIME TO FIRST TREATMENT ESCALATION | |
| | AND DRUG SURVIVAL) | 29 |
| | 8.2 Binary Endpoints | 29 |
| | 8.3 Continuous Endpoints | 29 |
| | 8.4 PATIENT REPORTED OUTCOMES (PROS) | 29 |
| 9 | STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES | 29 |
| | 9.1 Statistical methods | 29 |
| | 9.1.1 Analysis for Recurrent Event Data | 30 |
| | 9.1.2 Analysis for Time to Event Data | 31 |
| | 9.1.3 Analysis of Continuous Data | 31 |
| | 9.1.4 Analysis for Binary Data | 31 |
| | 9.1.5 Analysis of Categorical Data | 31 |
| | 9.1.6 Comparison between treatments | |
| | 9.2 Statistical Analyses | |
| | 9.2.1 Background and Demographic Characteristics and Study Disposition | 31 |
| | 9.2.2 Primary Analyses | |
| | 9.2.3 Secondary Analyses | |
| | 9.2.3.1 Time To First Treatment Escalation | |
| | 9.2.3.2 Rate of LDA | |
| | 9.2.3.3 Rate of Remission | |
| | 9.2.3.4 Change From Baseline in DAS28-4 (ESR) and DAS28-4 (CRP) | |
| | 9.2.3.5 Change from Baseline in Duration of Morning Stiffness | |
| | 9.2.3.6 Change from Baseline in FFbH | |
| | 9.2.3.7 Rate of Functional Remission | |
| | 9.2.3.8 Change from Baseline in EQ-5D | |
| | 9.2.3.9 Change from Baseline in FACIT-Fatigue | |
| Fi | nal Version 07-AUG-2023 | |

| | 9.2.3.10 Drug Survival Status of tofacitinib | 34 |
|----|--------------------------------------------------------------|----|
| | 9.2.3.11 Patient's Satisfaction with Drug treatment | |
| | 9.2.4 Safety Analyses | |
| | 9.2.5 Subgroup Analysis | |
| | 9.2.6 Summary of Analyses | |
| 10 | LIST OF TABLES AND TABLE SHELLS | 44 |
| 11 | REFERENCES | 44 |
| 12 | APPENDICES | 46 |
| 1 | 12.1 APPENDIX 1: DATA DERIVATION DETAILS | 46 |
| | 12.1.1 A1.1 Definition and use of visit windows in reporting | 46 |
| | 12.1.2 Definition of treatment escalations | |

### 1 LIST OF ABBREVIATIONS

| ACPA Anti-citrullinated protein antibodies ACR American Colleague of Rheumatology AE ALL All Patient Set BoMARD Biological Disease Modifying Antirheumatic Drug CAPEA COurse and Prognosis of Early Arthritis CDAI Clinical Disease Activity Index CI csDMARD Conventional Synthetic Disease Modifying Antirheumatic Drug CRF CRP C-reactive Protein DAS Disease Activity Score DMARD Disease Modifying Antirheumatic Drug EMA Disease Activity Score DMARD Disease Modifying Antirheumatic Drug EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFBH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid arthritis RF Rheumatoid arthritis RF Rheumatoid Thorapsis Set SAP Statistical Analysis Set SAP Statistical Analysis Set SAP Statistical Analysis Set SAS Safety Analysis Set SSO Swollen Joint Count SwpC SwmPC Supmars of Product Characteristics | Abbreviation | Definition |
|---|---|---|
| AE ALL All Patient Set ALL All Patient Set BDMARD Biological Disease Modifying Antirheumatic Drug CAPEA Course and Prognosis of Early Arthritis CDAI Clinical Disease Activity Index CI Confidence Interval csDMARD Conventional Synthetic Disease Modifying Antirheumatic Drug eCRF Electronic Case Report Form CRP C-reactive Protein DAS Disease Activity Score DMARD Disease Modifying Antirheumatic Drug EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFBH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PGA Patient Global Assessment of Arthritis RF Rheumatoid arthritis RF Rheumatoid arthritis RF Rheumatoid arthritis RF Rheumatoid arthritis SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SIC Swollen Joint Count | ACPA | Anti-citrullinated protein antibodies |
| ALL All Patient Set bDMARD Biological Disease Modifying Antirheumatic Drug CAPEA Course and Prognosis of Early Arthritis CDAI Clinical Disease Activity Index CI Confidence Interval Conventional Synthetic Disease Modifying Antirheumatic Drug eCRF Electronic Case Report Form CRP C-reactive Protein Case Report Form CRP DMARD Disease Modifying Antirheumatic Drug EMA European Medicines Agency EV-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFBH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RF Rheumatoid arthritis RF Rheumatoid arthritis RF Rheumatoid arthritis RF Rheumatoid arthritis RF Rheumatoid factor SAS Secondary Full Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SUC Swollen Joint Count | ACR | American Colleague of Rheumatology |
| bDMARD Biological Disease Modifying Antirheumatic Drug CAPEA Course and Prognosis of Early Arthritis CDAI Clinical Disease Activity Index CI Confidence Interval csDMARD Conventional Synthetic Disease Modifying Antirheumatic Drug eCRF Electronic Case Report Form CRP C-reactive Protein DAS Disease Activity Score DMARD Disease Modifying Antirheumatic Drug EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SIC Swollen Joint Count | AE | |
| CAPEA Course and Prognosis of Early Arthritis CDAI Clinical Disease Activity Index CI Confidence Interval csDMARD Conventional Synthetic Disease Modifying Antirheumatic Drug Antirheumatic Drug CCRF Electronic Case Report Form CRP C-reactive Protein DAS Disease Activity Score DMARD Disease Modifying Antirheumatic Drug EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Sct FFBH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Ra Rheumatoid arthritis RA Rheumatoid arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SWellen Joint Count | ALL | All Patient Set |
| CAPEA Course and Prognosis of Early Arthritis CDAI Clinical Disease Activity Index CI Confidence Interval csDMARD Conventional Synthetic Disease Modifying Antirheumatic Drug Antirheumatic Drug CCRF Electronic Case Report Form CRP C-reactive Protein DAS Disease Activity Score DMARD Disease Modifying Antirheumatic Drug EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Sct FFBH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Ra Rheumatoid arthritis RA Rheumatoid arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SWellen Joint Count | bDMARD | Biological Disease Modifying Antirheumatic Drug |
| CDAI Clinical Disease Activity Index CI Confidence Interval Conventional Synthetic Disease Modifying Antirheumatic Drug CCRF Electronic Case Report Form CRP C-reactive Protein DAS Disease Modifying Antirheumatic Drug EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis RA Rheumatoid arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAS Safety Analysis Set SIDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SGO Swollen Joint Count | CAPEA | |
| CI Confidence Interval csDMARD Conventional Synthetic Disease Modifying Antirheumatic Drug ECRF Electronic Case Report Form CRP C-reactive Protein DAS Disease Activity Score DMARD Disease Modifying Antirheumatic Drug EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Punctional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Rheumatoid arthritis RA Rheumatoid arthritis RF Rheumatoid arthritis RF Rheumatoid arthritis SAP Statistical Analysis Plan SAS Safety Analysis Set SIDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SIDC Swollen Joint Count | CDAI | |
| Antirheumatic Drug eCRF Electronic Case Report Form CRP C-reactive Protein DAS Disease Activity Score DMARD Disease Modifying Antirheumatic Drug EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PriGA Patient Global Assessment of Arthritis RA Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SIDAI Simplified Disease Activity Index SIGN Sovollen Joint Count | CI | |
| Antirheumatic Drug eCRF Electronic Case Report Form CRP C-reactive Protein DAS Disease Activity Score DMARD Disease Modifying Antirheumatic Drug EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PriGA Patient Global Assessment of Arthritis RA Rheumatoid factor SAE Scrious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SIDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SSIC Swollen Joint Count | csDMARD | Conventional Synthetic Disease Modifying |
| eCRF Creactive Protein DAS Disease Activity Score DMARD Disease Modifying Antirheumatic Drug EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SIC Swollen Joint Count | | |
| CRP C-reactive Protein DAS Disease Activity Score DMARD Disease Modifying Antirheumatic Drug EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SFAS Secondary Full Analysis Set SGAS Secondary Full Analysis Set | eCRF | |
| DMARD Disease Modifying Antirheumatic Drug EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | CRP | |
| DMARD Disease Modifying Antirheumatic Drug EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | DAS | Disease Activity Score |
| EMA European Medicines Agency EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | DMARD | |
| EQ-5D a self-report questionnaire (a quality of life instrument) developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FrbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | EMA | , , , |
| developed by the European Quality of Life (EuroQoL) Group ESR Erythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set | EO-5D | |
| ESR Eurythrocyte sedimentation rate EULAR European League Against Rheumatism EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SyJC Swollen Joint Count | | |
| EULAR EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | ESR | |
| EuroQoL European Quality of Life [Group] FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | EULAR | |
| FACIT Functional Assessment of Chronic Illness Therapy FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | EuroQoL | |
| FAS Full Analysis Set FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | | Functional Assessment of Chronic Illness Therapy |
| FFbH Functional Ability Questionnaire Hannover HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | FAS | |
| HCP Healthcare Professional JAK Januskinase LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | FFbH | |
| LDA Low disease activity MTX Methotrexate NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | НСР | |
| MTX NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | JAK | Januskinase |
| MTX NIS Non-Interventional Study PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | LDA | Low disease activity |
| PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | MTX | • |
| PF Prognostic Factor PhyGA Physician Global Assessment of Arthritis PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | NIS | Non-Interventional Study |
| PhyGAPhysician Global Assessment of ArthritisPPASPer Protocol Analysis SetPtGAPatient Global Assessment of ArthritisRARheumatoid arthritisRFRheumatoid factorSAESerious Adverse EventsSAPStatistical Analysis PlanSASSafety Analysis SetSDAISimplified Disease Activity IndexSFASSecondary Full Analysis SetSJCSwollen Joint Count | PF | |
| PPAS Per Protocol Analysis Set PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | PhyGA | |
| PtGA Patient Global Assessment of Arthritis RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | | · |
| RA Rheumatoid arthritis RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | | |
| RF Rheumatoid factor SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | | |
| SAE Serious Adverse Events SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | | |
| SAP Statistical Analysis Plan SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | | |
| SAS Safety Analysis Set SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | | |
| SDAI Simplified Disease Activity Index SFAS Secondary Full Analysis Set SJC Swollen Joint Count | | |
| SFAS Secondary Full Analysis Set SJC Swollen Joint Count | | |
| SJC Swollen Joint Count | | · |
| Din C Duninally of Floudet Characteristics | SmPC | Summary of Product Characteristics |

Final Version 07-AUG-2023 

TJC Tender Joint Count
TNFi Tumor necrosis factor inhibitor
tsDMARD Disease Modifying Antirheumatic Drug
VAS Visual Analogue Scale

2 AMENDMENTS FROM PREVIOUS VERSION(S)

The Protocol A3921302 ObservationalPlan Finalv1.1 23Aug2017.docx states that:

In order to collect comparable study data, visits 2 to 9 occurring +/- 14 days of the scheduled visit date will be used for data analysis.

As the visits will be scheduled according to clinical practice there are likely to be many visits outside of the windows defined in the protocol. To ensure the primary analysis incorporates all visits at which a patient might experience a treatment escalation all visits will be included. A further per-protocol analysis will be conducted using the analysis windows set out in Section 12.1.1.

Populations used during interim analyses were updated.

Additional details regarding the definition of the primary endpoint were added, because the definition provided in the protocol was not specific enough. Escalations were classified into 3 different types: Step-up, step-down or termination. The analysis of the primary endpoint will be conducted overall and per escalation type. A table with all possible treatment type changes has been added together with the corresponding type of escalation.

The assignment of escalations occurring in-between scheduled visits has been mostly aligned with that for the secondary endpoints for consistency across analyses and for greater precision of the assignment. In addition, imputation rules for missing values of covariates to be included in the analyses of the primary endpoint, have been added.

#### 3 INTRODUCTION

Note: in this document any text taken directly from the Non-Interventional (NI) study protocol is *italicised*.

Rheumatoid arthritis (RA) is a chronic autoimmune disease characterized by joint inflammation and destruction, progressive disability and adverse psychological effects.[1] Apart from musculoskeletal complications, RA patients suffer from increased frequencies and impacts of comorbidities such as cardiovascular and infectious diseases, osteoporosis or cancer, leading to higher mortality rates.[2,3,4] In addition, RA represents significant health and socioeconomic burdens for the individual patient and society, especially with regard to work disability and work productivity loss.[5,6]


·

With currently no curative therapy available, treatment strategies aim at controlling disease activity, alleviating signs and symptoms, maintaining physical function, improving quality of life, reducing the rate of joint damage, and, if possible, inducing complete remission.

Best treatment outcomes are achieved if RA is treated with disease modifying antirheumatic drugs (DMARDs) right from the beginning ('hit hard and early', 'window of opportunity'). [7,8,9,10] Furthermore, treatment strategies that aim at a predefined target ('treat-to-target' concept) have been shown to be superior to former, traditional approaches ('wait and see'). [11] Therefore, current European League Against Rheumatism (EULAR)-recommendations and the German S1 guideline derived from the EULAR-recommendations define treat-to-target as the basic therapeutic principle. The target to aim for is remission, especially in DMARD-naïve patients, or low disease activity, primarily in patients who failed previous therapies. [12] Although criteria for RA remission vary substantially in studies and clinical practice, the 28-joint Disease Activity Score (DAS28) is traditionally being widely used where DAS28 < 2,6 defines remission and DAS28  $\leq$  3,2 low disease activity. [13] According to EULAR recommendations, therapy has to be adjusted until the treatment target has been reached.

How is the treat to target approach applied in everyday care?

Despite insufficient response after 3 to 6 months therapy, treat-to-target recommendations of EULAR were only applied in 50% of the German course and prognosis of early arthritis cohort (CAPEA).[14] In an analysis of a cohort from the "Kerndokumentation", a national database of the German Collaborative Arthritis Centres, 45% of patients were not within DAS28 low disease activity range and therefore would have needed adaption of therapy according to current treatment guidelines. In contrast, rheumatologists' global assessment of disease activity differed, 80% perceived their patients to be in the low disease activity range and, hence, as being adequately treated.[15]

These observations suggest that in a real-world setting, criteria other than calculated DAS28 remission or low disease activity alone may guide treatment decisions. Among such criteria, satisfaction with drug treatment is of particular interest. On the one hand, a patient who is content with his current therapy is less likely to be willing to change a therapy solely to achieve a better DAS28 score. On the other hand, patient preference and satisfaction of a therapy strongly affects adherence to a prescribed medication, ultimately affecting treatment outcome and efficacy. A factor known to impact on patient satisfaction with a prescribed treatment is the route of administration. Here, several studies point to a preference for oral therapies, also among second-line DMARDs.[16,17]

Recently, tofacitinib, an orally applied DMARD of the new class called Janus-Kinase-Inhibitors (JAK-Inhibitors) has been brought into the market in the European Union. tofacitinib is indicated in combination with methotrexate (MTX) for the treatment of moderate to severe active rheumatoid arthritis (RA) in adult patients who have responded inadequately to, or who are intolerant to one or more DMARD. Due to oral administration


oftofacitinib, the impact of patient's satisfaction with drug treatment on therapy decisions by rheumatologists may be especially pronounced.

EULAR recommendations have now endorsed individual patient related factors such as patient preferences and comorbidities as an overarching principle in the management of RA.

#### 3.1 STUDY DESIGN

This is a 60-month, prospective, non-interventional, multi-centre study to evaluate the impact of the following factors on the number of treatment escalations of tofacitinib patients in 24 months.

Eligible patients will be followed up from the date of first tofacitinib prescription for 24 months. Patients who are switched from the initial tofacitinib therapy to other therapies will also be followed up to 24 months. Patient documentation is expected quarterly as per standard clinical practice.

This study observes drug prescription and follow-up visits in daily medical care. Therapeutic strategies and frequency of patient follow-up are decided by the treating physician.

Figure 1. Study Design



The planned recruitment period is 36 months. With planned observation duration of 24 months per patient, the entire study would thus last for 60 months. The study started in October 2017 and, due to an extension of the recruitment period of 9 months, the study will end in July 2023. Overall, about 1500 patients in about 200 centres in Germany are to be included in this non-interventional study.


The schedule of activities table provides an overview of the visits that may be documented. Refer to the STUDY PROCEDURES and ASSESSMENTS sections of the protocol for detailed information on each documentation and assessment.

According to his clinical practice the HCP may schedule visits (unplanned visits) in addition to those listed on the schedule of activities, in order to conduct evaluations or assessments required to protect the well-being of the patient. As this is a non-interventional study none of these visits are mandatory and every visit should be scheduled according to clinical practice.


**Table 1. Schedule of Activities** 

| Study Week | Baseline<br>(Enrolmen() | Month 3 | Month 6 | Month<br>9 | Month<br>12 | Month<br>15 | Month<br>18 | Month<br>21 | Month<br>24 |
|---|---|---|---|---|---|---|---|---|---|
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| Info1med Consent | х | | | | | | | | |
| Initial dia211osis of RA | х | | | | | | | | |
| Proimostic factors | X | | | | | | | | |
| Relevant comorbidities | X | | | | | | | | |
| Demographic data | Х | | | | | | | | |
| Insurance type | х | | | | | | | | |
| Smoking history and cwTent smoking status | Х | | | | | | | | |
| Physical Examination (weight, height) | Х | | | | | | | | |
| Inclusion/Exclusion criteria | х | | | | | | | | |
| Varicella vaccination status | х | | | | | | | | |
| Prior drug treatment of RA | Х | | | | | | | | |
| RA-treatment with tofacitinib and/or other DMARDs | Х | Х | х | х | Х | х | Х | Х | х |
| Concomitant treatment of RA with Glucocorticoids | х | х | х | х | Х | х | х | х | х |
| InflammatoIY Markers | Χ | Х | Х | Х | Х | Х | Х | Х | Х |
| Documentation of AE | х | х | х | х | Х | х | х | х | х |
| Number of swollen and tender joints | х | х | х | х | Х | Х | х | х | Х |
| Duration of Moming stiffness | X | Х | Х | Х | Х | Х | X | Х | Х |
| Patient's Global Assessment of<br>Arthritis | х | х | х | х | Х | х | х | х | х |
| Physician's Global Assessment of Arthritis | х | х | х | х | Х | х | х | х | х |
| Patient's Assessment of Arthritis Pain | Χ | X | х | Х | Х | Х | X | X | Х |
| Functional Ability Questionnaire<br>Hannover (FFbH) | х | х | х | х | Х | х | х | х | х |
| EuroOoL E0-5D-3L | Х | Х | х | Х | Х | Х | X | Х | Х |
| FACIT- Fatigue Scale | Х | Х | х | Х | Х | Х | Х | Х | Х |
| Patient's satisfaction with diug treatment | х | х | х | х | X | х | х | х | x |

#### **3.2 STUDY POPULATION**

Patients attending can be included by the HCP if they fulfil all selection criteria for the study and are started on treatment with tofacitinib for moderate to severely active rheumatoid arthritis.

All visits shall be scheduled according to clinical practice. The treatment of a patient is independent from the patient enrolment into the study. Within this study 9 visits may be documented. At each visit patients will undergo procedures in compliance with the country


*label and as per standard of care.* The protocol states that data from Visits 2 to 9 occurring +/- 14 days of the scheduled visit date will be used for the analysis, however this definition will be amended within the SAP (see Sections 12.1.1 and 6 for further detail).

After a training session the sites will get access to the eCRF, where the data and findings of the patient are documented. Additionally, a folder with questionnaires will be provided. The collection of all data is prospective.

Dose and duration of treatment should be based on clinical and individual needs and are determined by the treating physician. To provide accurate information regarding the treatment, the initial tofacitinib dose and all changes and the reasons for changes are documented during the course of the evaluation. The concomitant treatment of rheumatoid arthritis with Glucocorticoids is determined by the treating physician and is registered in the documentation sheet.

#### 3.2.1 TREATMENT/COHORT LABELS

For the primary analysis, the number and timing of treatment escalations of tofacitinib patients in 24 months will be presented (see Section 7.1.1). The treatment labels for other analyses are presented below:

#### 3.2.1.1 TREATMENT LABEL FOR SECONDARY ANALYSIS

tofacitinib (in Monotherapy or in Combination with MTX)

## 3.2.1.2 TREATMENT LABEL FOR SECONDARY ANALYSIS – SUBGROUP SEQUENCE OF THERAPY

tofacitinib in Monotherapy
tofacitinib in Monotherapy → Combination with MTX
tofacitinib in Combination with MTX
tofacitinib in Combination with MTX → tofacitinib Monotherapy

#### 3.3 STUDY OBJECTIVES

The objective of this non-interventional study is to identify key factors that are driving treatment decisions by rheumatologists in the treatment of RA patients starting treatment with tofacitinib in a real world setting. In addition to DAS28 score, following factors may play an important role: difference between DAS28 at start of therapy and after 3-6 months, physician's global assessment of disease activity, patients' global assessment of disease activity, arthritis pain and patient's overall satisfaction with treatment.


#### 4 INTERIM AND FINAL ANALYSES

#### 4.1 INTERIM ANALYSIS

A first interim analysis was carried out after 50% of the planned number of patients (i.e. 750 patients) had reached their M12 visit. The M12 interim analysis only considered the secondary endpoints.

Two analysis populations were used:

- 1) M12 Population: all those patients that have completed the M12 visit
- 2) Baseline Population: all those that have completed at least the baseline visit.

A second interim analysis was carried out after 50% of patients had reached their M24 visit. The M24 interim analysis considered the secondary endpoints in addition to summary tables of the primary endpoint (no statistical modelling was undertaken within the interim analysis). Two analysis populations were used:

- 1) M24 Population Set: all those patients that have completed the M24 visit
- 2) M12 Population Set: all those patients that have completed the M12 visit
- 3) Baseline Population Set: all those that have completed at least the baseline visit.

A third Interim Analysis was conducted with a database export of 31<sup>st</sup> January 2022 following the methods of the second Interim Analysis described above.

The outputs required for the interim analyses were a subset of the final outputs and methods were the same as for the final analysis. Therefore, a separate analysis plan was not required. Details of the output requirements were provided in the list of tables.

#### 4.2 FINAL ANALYSIS

The final analysis will include all enrolled patients and will be carried out after all patients have reached their final visit (at month 24). The final datasets will be extracted from the database and locked before final analysis. Any exclusions from the analysis will be agreed and documented prior to database lock. The final analysis will be based on the populations described under 6 Analysis Sets/ populations, the populations M12 and M24 used for the interim analyses will not be used for the final analysis.

#### 4.3 POOLED ANALYSIS

The data from this protocol is also planned to be included in a pooled analysis with other European non-interventional studies. Details will be included in a separate analysis plan. The pooled analysis is not part of the final analysis.


#### 5 HYPOTHESES AND DECISION RULES

Data will be summarised descriptively. Tables will include appropriate confidence intervals (CIs) so as to provide information on the precision of the estimates. For the primary endpoint a predictive model will be used to assess the impact of a number of factors on the number and timing of treatment escalations.

#### 6 ANALYSIS SETS/ POPULATIONS

#### 6.1 ALL PATIENT SET

The All Patient Set (ALL) includes all patients enrolled in the study and will include all data collected at both scheduled and unscheduled visits. The ALL will primarily be used for disposition analyses and listings.

#### 6.2 FULL ANALYSIS SET

The Full Analysis Set (FAS) will include all patients who receive at least one dose of tofacitinib and have at least one post-baseline visit. The primary analysis will use the FAS. The FAS will include all data collected during the study, both scheduled and unscheduled visits.

The protocol states that patients will be enrolled if they fulfil all selection criteria for the study and are started on treatment with tofacitinib for moderate to severely active rheumatoid arthritis.

#### 6.3 SECONDARY FULL ANALYSIS SET

Patients with data collected while taking tofacitinib will be assigned to the Secondary Full Analysis Set (SFAS) at a given time point, which will be used for all secondary endpoint analyses. A patient is considered on tofacitinib at a given timepoint if the patient has not terminated or paused tofacitinib at the time of the visit or event. Termination or pauses are documented in eCRF instrument "Rheumatologische Medikation" for therapy class tsDMARD/bDMARD, where variable *Change* (BDCM.CHANGECD) is set to "Therapy stop" = termination or set to "Therapy paused" = pause.

#### 6.4 SAFETY ANALYSIS SET

The Safety Analysis Set (SAS) will consist of all patients who receive at least one dose of tofacitinib. All reporting of safety data will utilize the SAS.

#### 6.5 PER PROTOCOL ANALYSIS SET


Patients with data collected at scheduled visits, which fall within the defined visit windows (see section 12.1.1) will be assigned to the Per-Protocol Analysis Set (PPAS).

#### 6.6 SUBGROUPS

The following subgroups will be considered for the analysis of the secondary endpoints if sufficient numbers of patients are available.

- 1) Sequence of therapy, where subgroups (with treatment labels as defined in 2.2.1.2) are:
  - a) Patients who were on tofacitinib as a Monotherapy throughout the study.
  - b) Patients who were on tofacitinib as a Monotherapy and switched to tofacitinib in combination with MTX.
  - c) Patients who were on tofacitinib in Combination with MTX throughout the study.
  - d) Patients who started on tofacitinib in Combination with MTX and switched to tofacitinib as a Monotherapy.

Note: Only a patient's first switch will be used to classify them into a subgroup.

If above classification is too granular, the following subgroups will be used for sequence of therapy:

- a) Patients who were on tofacitinib as a Monotherapy throughout at least 60% of their observational time
- b) Patients who were on tofacitinib as a Combination with MTX throughout at least 60% of their observational time
- 2) Medication history of RA treatment where the subgroups are:
  - a) Those on 2<sup>nd</sup> line treatments prior to starting study.
  - b) Those on 3<sup>rd</sup> line treatments prior to starting study.

The eCRF will be referred to for a list of drug names for each category.

- 3) Patient's Switch Status, where the subgroups are:
  - a. Patients with a treatment step- up as defined in section 7.1.1: switch up
  - b. Patients that remain on tofacitinib treatment or patients with a treatment step-down: no switch up
- 4) Number of Treatment Escalations (as defined in section 7.1.1):
  - a) Patients with no treatment escalations.


- b) Patients with 1 treatment escalation.
- c) Patients with 2 treatment escalations.
- d) Patients with 3 or more treatment escalations.

#### 7 ENDPOINTS AND COVARIATES

#### 7.1 EFFICACY/EFFECTIVENESS ENDPOINT(S)

#### 7.1.1 PRIMARY ENDPOINTS

Number and timing of treatment escalations of tofacitinib patients in 24 months, where Treatment Escalation in this study is defined as a switch to another DMARD or combination of DMARDs when compared to the last visit.

The following types of escalations will be distinguished:

- 1. Treatment **Termination**, which is the termination of a DMARD (or multiple when on combination therapy) without starting a new DMARD therapy. Premature study terminations (without documented treatment termination) will not be considered treatment terminations.
- 2. Treatment **Step-up** which is an increase from the current treatment regime towards e.g. a combination of DMARDs
- 3. Treatment **Step-down**, which is a de-escalation from the current treatment regime, e.g. from combination therapy to monotherapy

Patients start their therapy at baseline with tofacitinib either in Monotherapy or in Combination therapy with MTX. Subsequent therapy changes are documented on eCRF instrument "Rheumatologische Medikation" by:

- adding additional DMARDs on top of the current therapy
- stopping the current DMARD in monotherapy and adding a new DMARD
- stopping one of multiple DMARDs when on combination therapy
- stopping one of multiple DMARDs when on combination therapy and adding a new DMARD
- stopping all DMARDs and not starting a new therapy. The escalation types depend on the combination of DMARD classes (tsDMARD vs bDMARD vs TNFi vs csDMARD). The eCRF does not explicitly distinguish between tsDMARD vs bDMARD vs TNFi, but combines all rheumatic medications belonging to the above classes under


tsDMARD/bDMARD. For the definition of treatment escalations, the following assignment of rheumatic medication to DMARD classes will be done:

#### tsDMARDS:

- baricitinib
- upadacitinib
- filgotinib

#### TNFi:

- etanercept
- adalimumab
- certolizumab
- golimumab
- infliximab

#### bDMARDs (excluding TNFi):

- abatacept
- rituximab
- anakinra
- tocilizumab
- sarilumab

For details of treatment escalations, e.g., which DMARD class addition or reduction leads to a particular escalation type, see table 12.2 in section 12.1.2.

#### 7.1.2 SECONDARY ENDPOINTS

This study has a number of secondary efficacy endpoints:

#### 7.1.2.1 TIME TO FIRST TREATMENT ESCALATION

For patients who experience a treatment step-up (as defined in section 7.1.1), the Treatment Escalation Status and Time to First Treatment Escalation will be recorded as follows:

- Status = 1
- Time = Date of first treatment escalation Date of initiation on tofacitinib

For patients who don't experience a treatment escalation, the Treatment Escalation Status and time to first treatment escalation will be recorded as follows:

• Status = 0


• Time = Date of final visit – Date of initiation on tofacitinib

If a patient is lost to follow-up or withdraws from the study, they will be censored at the date of their last visit.

The analysis for time to first treatment escalation type step-up may be extended to escalation type step-down.

#### **7.1.2.2 RATE OF LDA**

The Rate of Low Disease Activity (LDA) will be calculated over time for patients taking tofacitinib using 4 different definitions:

- a) SDAI  $\leq$  11;
- b) CDAI ≤10;
- c) DAS 28-4 (ESR)  $\leq$  3.2 and
- d) DAS 28-4 (CRP)  $\leq$  3.2.

These are defined in detail below.

#### 7.1.2.2.1 SDAI LDA

At each time point (M3, M6, M9, M12, M15, M18, M21, M24) SDAI LDA is derived as:

SDAI\_LDA = 1 if SDAI 
$$\leq$$
 11 SDAI LDA = 0, otherwise.

The proportion of patients in SDAI LDA at Month X is then calculated as:

No. of patients with SDAI LDA at Month X / Total Number of patients with non-missing SDAI LDA at Month X.

#### 7.1.2.2.2 CDAI LDA

At each time point (M3, M6, M9, M12, M15, M18, M21, M24) CDAI LDA is derived as:

CDAI\_LDA = 1 if 
$$CDAI \le 10$$
  
CDAI\_LDA = 0, otherwise.

The proportion of patients in CDAI LDA at Month X is then calculated as:

No. of patients with CDAI LDA at Month X / Total Number of patients with non-missing CDAI LDA at Month X.


### 7.1.2.2.3 DAS28-4 (ESR) LDA

At each time point (M3, M6, M9, M12, M15, M18, M21, M24) DAS 28-4 (ESR) LDA is derived as:

```
DAS 28-4 (ESR) LDA = 1 if DAS 28-4 (ESR) \leq 3.2. DAS 28-4 (ESR) LDA = 0, otherwise.
```

DAS28-4 (ESR) is calculated as in Section 7.1.2.4.1

The proportion of patients in DAS 28-4 (ESR) LDA at Month X is then calculated as:

No. of patients with DAS 28-4 (ESR) LDA at Month X / Total Number of patients with non-missing DAS 28-4 (ESR) LDA at Month X.

#### 7.1.2.2.4 DAS28-4 (CRP) LDA

At each time point (M3, M6, M9, M12, M15, M18, M21, M24) DAS 28-4 (CRP) LDA is derived as:

DAS 28-4 (CRP)\_LDA = 1 if DAS 28-4 (CRP) 
$$\leq$$
 3.2. DAS 28-4 (CRP) LDA = 0, otherwise.

DAS28-4 (CRP) is calculated as in Section 7.1.2.4.1

The proportion of patients in DAS 28-4 (CRP) LDA at Month X is then calculated as:

No. of patients with DAS 28-4 (CRP) LDA at Month X / Total Number of patients with non-missing DAS 28-4 (CRP) LDA at Month X.

#### 7.1.2.3 RATE OF REMISSION

The Rate of Remission will be calculated over time for patients taking to facitinib, using 5 definitions:

- a) American College of Rheumatology (ACR) European League Against Rheumatism (EULAR) Boolean remission criteria;
- b) Simplified Disease Activity Index (SDAI)  $\leq 3.3$ ;
- c) Clinical Disease Activity Index (CDAI) ≤2.8;
- d) DAS 28-4 (ESR)  $\leq$  2.6 and
- e) DAS28-4 (CRP) < 2.6


These are defined in more detail below.

#### 7.1.2.3.1 ACR-EULAR BOOLEAN REMISSION CRITERIA

At each time point (M3, M6, M9, M12, M15, M18, M21, M24) ACR Remission is derived as:

ACR Remission = 1, if:  $SJC28 \le 1$ ,  $TJC28 \le 1$ ,  $CRP \le 1$  mg/dL, and  $PtGA \le 2$ cm

ACR Remission = 0, Otherwise.

The proportion of patients in ACR Remission at Month X is then calculated as:

No. of patients with ACR Remission at Month X / Total Number of patients with non-missing ACR Remission at Month X.

#### 7.1.2.3.2 SDAI REMISSION

At each time point (M3, M6, M9, M12, M15, M18, M21, M24) SDAI is calculated as:

SDAI = TJC28 + SJC28 + PhyGA in cm + PtGA in cm + CRP in mg/dL

SDAI\_Remission = 1, if SDAI  $\leq 3.3$ SDAI\_Remission = 0, otherwise.

The proportion of patients in SDAI Remission at Month X is then calculated as:

No. of patients with SDAI Remission at Month X / Total Number of patients with non-missing SDAI Remission at Month X.

#### 7.1.2.3.3 CDAI REMISSION

At each time point (M3, M6, M9, M12, M115, M18, M21, M24) CDAI Remission is derived as:

CDAI = TJC28 + SJC28 + PhyGA in cm + PtGA in cm

CDAI\_Remission = 1, if CDAI  $\leq 2.8$ CDAI\_Remission = 0, otherwise.

The proportion of patients in CDAI Remission at Month X is then calculated as:

No. of patients with CDAI Remission at Month X / Total Number of patients with non-missing CDAI Remission at Month X.


#### 7.1.2.3.4 DAS28-4 (ESR) REMISSION

At each time point (M3, M6, M9, M12, M115, M18, M21, M24) DAS 28-4 (ESR) Remission is derived as:

DAS 28-4 (ESR)\_Remission = 1, if DAS28-4 (ESR) 
$$\leq$$
 2.6 DAS 28-4 (ESR) Remission = 0, otherwise.

The proportion of patients in DAS 28-4 (ESR) Remission at Month X is then calculated as:

No. of patients with DAS 28-4 (ESR) Remission at Month X / Total Number of patients with non-missing DAS 28-4 (ESR) Remission at Month X.

#### 7.1.2.3.5 DAS28-4 (CRP) REMISSION

At each time point (M3, M6, M9, M12, M115, M18, M21, M24) DAS 28-4 (CRP) Remission is derived as:

```
DAS 28-4 (CRP)_Remission = 1, if DAS28-4 (CRP) \leq 2.6 DAS 28-4 (CRP) Remission = 0, otherwise.
```

The proportion of patients in DAS 28-4 (CRP) Remission at Month X is then calculated as:

No. of patients with DAS 28-4 (CRP) Remission at Month X / Total Number of patients with non-missing DAS 28-4 (CRP) Remission at Month X.

#### 7.1.2.4 CHANGE FROM BASELINE IN DAS28-4 (ESR) AND DAS28-4 (CRP)

#### 7.1.2.4.1 DAS28-4

DAS28-4 (ESR) =  $0.56*\sqrt{\text{TJC28}} + 0.28*\sqrt{\text{SJC28}} + 0.70*\text{In(ESR in mm/ hour)} + 0.014*\text{PtGA in mm}$ .

DAS28-4 (CRP) is similarly calculated by:

DAS28-4 (CRP) = 
$$0.56*\sqrt{\text{TJC28}} + 0.28*\sqrt{\text{SJC28}} + 0.36*\ln(\text{CRP in mg/l} + 1) + 0.014*\text{PtGA in mm} + 0.96$$

Where TJC28 is the Tender Joint Count, SJC28 is the Swollen Joint Count, CRP is the Creactive protein in mg/L, ESR is the Erythrocyte Sedimentation Rate in mm/first hour and


PtGA is the Patient's Global Assessment of Health in mm. PtGA will be used in this calculation.

The change from baseline in DAS28-4 (ESR) will be calculated at each time point as:

DAS28-4 (ESR) at time point – DAS28-4 (ESR) at baseline.

Similarly change from baseline in DAS28-4 (CRP) will be calculated at each time point as:

DAS28-4 (CRP) at time point – DAS28-4 (CRP) at baseline.

Change from Baseline in DAS 28-4 at all time points (M3, M6, M9, M12, M15, M18, M21, M24) will be presented.

#### 7.1.2.5 CHANGE FROM BASELINE IN DURATION OF MORNING STIFFNESS

The duration of stiffness in the morning will be provided in the eCRF.

The change from baseline in duration of morning stiffness will be calculated as.

Morning Stiffness at time point – Morning Stiffness at baseline.

#### 7.1.2.6 CHANGE FROM BASELINE IN FFBH

The FFbH questionnaire consists of 18 questions with 3 possible responses (Yes; Yes, but with effort; No or only with outside help).

The total score is the sum of the scores of all 18 questions, where for each question:

- Yes = 2 points
- Yes, but with effort = 1 point
- No or only with outside help = 0 points

The Functional capacity [%] is then

(Total score\*100)/(2\*number of valid responses)

The change from baseline will then be calculated at each time point as:

Functional capacity at timepoint – Functional capacity at baseline

Change from Baseline in FFbH functional capacity at all time points (M3, M6, M9, M12, M115, M18, M21, M24) will be presented.


#### 7.1.2.7 RATE OF FUNCTIONAL REMISSION (FFBH)

At each time point FFbH remission is derived as:

FFbH Remission = 1, if FFbH > 83%

FFbH Remission = 0, Otherwise

The proportion of patients with FFbH Functional Remission at Month X is then calculated as:

No. of patients with FFbH\_Remission at Month X / Total Number of patients with non-missing FFbH Remission at Month X.

#### 7.1.2.8 CHANGE FROM BASELINE IN EQ-5D

The EQ-5D is a self-reported questionnaire developed by the European Quality of Life (EuroQoL) Group. It is a standardised instrument used to measure quality of life. Change from baseline in EQ-5D will be collected over time and analysed for patients taking tofacitinib. It is based on five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three responses and the patient is asked to select the response that best describes them. The responses are scored 1-3 as shown in Table 2.

Table 2: EQ-5D scores

| Dimension | Response | Score |
|---|---|---|
| Mobility | I have no problems in walking about | 1 |
| | I have some problems in walking about | 2 |
| | I am confined to bed | 3 |
| Self-care | I have no problems with self-care | 1 |
| | I have some problems washing or dressing myself | 2 |
| | I am unable to wash or dress myself | |
| Usual activities (e.g. | I have no problems with performing my usual | |
| work, study, | activities | |
| housework, family or | I have some problems with performing my usual 2 | |
| leisure activities) | activities | |
| | I am unable to perform my usual activities | 3 |
| Pain/discomfort | I have no pain or discomfort | |
| | I have moderate pain or discomfort | 2 |
| | I have extreme pain or discomfort | 3 |


| Anxiety/depression | I am not anxious or depressed | 1 |
|--------------------|--------------------------------------|---|
| | I am moderately anxious or depressed | 2 |
| | I am extremely anxious or depressed | 3 |

The score for each dimension is weighted in accordance with **Table 3**.

**Table 3: EQ-5D Weightings** 

Weights from Germany are used:

| <b>EQ-5D Dimension</b> | Score = 1 | Score = 2 | Score = 3 |
|------------------------|-----------|-----------|-----------|
| Mobility | 0 | 0.069 | 0.314 |
| Self-Care | 0 | 0.104 | 0.214 |
| Usual Activities | 0 | 0.036 | 0.094 |
| Pain/Discomfort | 0 | 0.123 | 0.386 |
| Anxiety/Depression | 0 | 0.071 | 0.236 |

The following algorithm is then applied to calculate the EQ-5D Total Score:

- 1. If all five EQ-5D dimensions have a score of 1 then the EQ-5D Total Score is 1.
- 2. If any of the five EQ-5D dimensions have a score of 3, then the EQ-5D Total Score is:

$$1 - 0.081 - (\sum_{1} weighted dimension score) - 0.269$$

3. If none of the five EQ-5D dimensions has a score of 3, then the EQ-5D Total Score is:

$$1 - 0.081 - (\sum_{i=1}^{5} weighted dimension score)$$

Missing weighted dimension scores are replaced by the mean of the non-missing weighted dimension scores. If a weighted score is missing and replaced in this way by a mean weighted score of zero, step 3 of the algorithm is applied.

The change from baseline in EQ-5D will be calculated for each time point as:

EQ-5D at timepoint 
$$X - EQ-5D$$
 at baseline


#### 7.1.2.9 CHANGE FROM BASELINE IN FACIT-FATIGUE

The FACIT-Fatigue score is derived by taking the sum of the scores for the 13 questions in the instrument, resulting in a score between 0 and 52.

The change from baseline in FACIT-Fatigue score will be calculated for each time point as:

FACIT-Fatigue score at time point X – FACIT-Fatigue score at baseline

#### 7.1.2.10 DRUG SURVIVAL STATUS OF TOFACITINIB

For patients who terminate tofacitinib, the drug survival status will be recorded as follows:

Those who terminate tofacitinib:

- Status = 1
- Time = Termination date to facitinib Date of initiation on to facitinib

Tofacitinib is terminated when indicated on instrument "Rheumatologische Medikation" for therapy class tsDMARD/bDMARD variable *Change* (BDCM.CHANGECD) is set to "Therapy stop". Tofacitinib pauses, where variable *Change* is set to "Therapy paused", are not considered terminations.

Patients who do not terminate tofacitinib:

- Status = 0
- Time = Date of final visit Date of initiation on tofacitinib

If patient is lost to follow-up or withdraws from the study they will be censored at the date of their last visit.

#### 7.1.2.11 PATIENT'S SATISFACTION WITH DRUG TREATMENT

Patient's overall satisfaction with treatment is assessed via a 5-point likert question (extremely dissatisfied, dissatisfied, neither satisfied nor dissatisfied, satisfied and extremely satisfied).


At each visit, Visit X, overall satisfaction will be presented only for those who remained on tofacitinib at the last visit, Visit X-1. This will be split by those who stop taking tofacitinib at Visit X and those that remain on tofacitinib at Visit X.

#### 7.2 SAFETY ENDPOINTS

Incidence and severity of all adverse events including serious adverse events (SAEs).

The reporting of safety data will be in accordance with Pfizer Data Standards.

#### 7.3 COVARIATES, FACTORS AND POTENTIAL CONFOUNDERS

#### 7.3.1 FACTORS OF INTEREST FOR PRIMARY ANALYSIS

The following covariates will be included in the primary analysis:

- a. DAS 28-4 (ESR) LDA (see sections 6.1.2.4.1 and 6.1.2.2.3 for derivations) [Note: this is a binary endpoint].
- b. Indicator variable for whether patient has achieved change from baseline of DAS28-4 (ESR) > 1.8 (see section 6.1.2.4.1 for derivations of DAS28-4 (ESR)) [Note: this is a binary endpoint].

Change from baseline will be calculated as:

 $\Delta DAS28-4$  (ESR) = DAS28-4 (ESR) at time point – DAS28-4 (ESR) at baseline

If a patient has achieved  $\Delta DAS28-4$  (ESR) > 1.8 the indicator will be 1,

If  $\Delta DAS28-4$  (ESR) > 1.8 is not achieved, the indicator will be 0.

- c. Physician Global Assessment of Arthritis measured on a visual analogue scale (0-100mm).
- d. Patient's Global Assessment of Arthritis measured on a visual analogue scale (0-100mm).
- e. Patient's Assessment of Arthritis Pain measured on a visual analogue scale (0-100mm).
- f. Patient's overall satisfaction with treatment:


For each patient the response to the question 'How satisfied are you with the drugs that you have received for your arthritis since your last visit?' will be assigned as below:

- 0 = extremely dissatisfied,
- 1= dissatisfied,
- 2 = neither satisfied nor dissatisfied,
- 3 = satisfied
- 4 = extremely satisfied

### 7.3.2 FACTORS OF INTEREST FOR SENSITIVITY OF THE PRIMARY ANALYSIS

The following covariates will be included in a sensitivity analysis of the primary endpoint:

- a. DAS28-4 with Erythrocyte Sedimentation Rate (ESR) (section 7.1.2.4.1). [Note: this is a continuous endpoint].
- b. ΔDAS28-4 (ESR), [Note: this is a continuous endpoint].
- c. Physician Global Assessment of Arthritis
- d. Patient's Global Assessment of Arthritis
- e. Patient's Assessment of Arthritis Pain
- f. Patient's overall satisfaction with treatment
- g. Incidence of comorbidities
  - o 1 if patient has at least one comorbidity
  - o 0 if no comorbidities are recorded

### 7.3.3 POTENTIAL CONFOUNDERS TO BE INCLUDED IN THE PRIMARY ANALYSIS


A number of potential confounders will also be included in the primary analysis and all sensitivity analyses:

- Age at baseline
- Gender
- Duration of disease at baseline
- Indicator of tofacitinib dose
  - o 1 if recommended dose of 5mg per day (i.e. TofInterval = BID),
  - o 0 if reduced dose of 2.5mg per day (i.e. TofInterval = Daily).
- Poor prognostic factors (PF) indicator (1 if at least one Poor PF is present, 0 otherwise)
- Indicator of dose of MTX or combination partner (1 if increase in dose since last visit, 0 otherwise)
- Indicator of dose of Glucocorticoids (1 if increase in dose since last visit, 0 otherwise)
- Whether patient on 2<sup>nd</sup> or 3<sup>rd</sup> line treatment (see below)

A patient is defined as on 2<sup>nd</sup> line treatment if they were prescribed only csDMARDs prior to enrolling in the study.

A patient is defined as on 3<sup>rd</sup> line treatment if they were prescribed bDMARDs prior to enrolling in the study.

For a list of the medications considered to be csDMARDs and bDMARDs please see the eCRF.

- Indicator of tolerability issues (1 if treatment termination due to tolerability issues, 0 otherwise).
- Indicator of efficacy issues (1 if treatment termination due to efficacy issues, 0 otherwise).
- Incidence of the following comorbidities documented at the baseline visit (a term will be fitted for each comorbidity with the value 1 if the comorbidity is recorded for a patient or 0 otherwise):
  - o Ischemic cardiovascular disease
  - o Malignancies
  - o Infections
  - o Gastro disease
  - Osteoporosis
  - Depression

Any other variables observed to be potential confounders will also be investigated.


#### 8 HANDLING OF MISSING VALUES

# 8.1 TIME TO EVENT (PRIMARY ANALYSIS, TIME TO FIRST TREATMENT ESCALATION AND DRUG SURVIVAL)

Time to event should be determined for the events without any date imputation.

If a patient experiences the event of interest the status will be 1, and the time will be the time at which the event occurred (or visit at which it was recorded).

If a patient doesn't experience the event of interest the status will be 0, and the time will be the last time that the patient was known to be in the study (last visit). If this is not the end of the study then the time will be censored at this time point.

The primary endpoint is a time-to-event endpoint, although it takes into account the possibility of multiple events occurring for each patient. For each patient the data for analysis should consist of the times at which they experienced the event of interest and the values of the covariates at each time point. Any missing data within the covariates to be included in the models for primary analysis will be replaced by the nearest available value to the event. If more than one value qualifies, the later value will be used .

#### 8.2 BINARY ENDPOINTS

Missing data will not be imputed unless stated otherwise.

#### 8.3 CONTINUOUS ENDPOINTS

Missing data will not be imputed unless stated otherwise.

#### 8.4 PATIENT REPORTED OUTCOMES (PROS)

The questionnaires that will be used in the study (EQ-5D-5L, FACIT-Fatigue and FFbH) are accompanied by rules for replacing missing values. If these rules result in the patient having a missing score at a visit, then the missing values will be assumed to be missing at random.

#### 9 STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES

#### 9.1 STATISTICAL METHODS


Descriptive statistics will be presented to describe patient characteristics. Generally, categorical covariates will be described by frequency distribution while continuous covariates expressed in terms of their mean and standard deviation or median and interquartile range (IQR) as appropriate. Graphical displays may also be used.

#### 9.1.1 ANALYSIS FOR RECURRENT EVENT DATA

In order to account for the possibility that there are multiple events occurring for each patient cox-proportional hazards modeling will be used with adjustment for recurrent events. This involves fitting either the Andersen and Gill or Prentice, Williams and Peterson gap-time models to the data.

For each patient, the data will be split into time periods, then data for each time window should include the patient's status, the time of event (if the event occurred) and the value of each of the factors of interest:

So, for patient A, who had events at M6 and M18, their data could look like this:

| Patient | Start | Stop | Treatment | Factor A | Factor B | Factor C |
|---------|-------|------|------------|----------|----------|----------|
| | | | Escalation | | | |
| | | | Status | | | |
| A | 0 | M6 | 1 | 3.9 | 0.6 | -10 |
| A | M6 | M12 | 0 | 3.0 | 1.5 | -20 |
| A | M12 | M8 | 1 | 2.8 | 1.7 | -10 |
| A | M18 | M24 | 0 | 2.2 | 2.3 | -10 |

The cox proportional hazards model (using PROC PHREG) is then used, including the factors of interest (Section 7.3.1) to determine which, if any of them, have an impact on the rate at which treatment changes occur.

Any potential confounders should be included in the model also (Section 7.3.3).

The estimated event rate will be presented, along with 95% confidence interval and p-value, for each of the covariates of interest. Note: These will not be presented for the variables considered to be confounders.

The number and proportion of people experiencing an event at each time point will be presented.

Supportive tables will also be presented which summarises each of the covariates in the model at each visit.

The analysis will be performed for each type of escalation as defined in section 7.1.1 and overall.


#### 9.1.2 ANALYSIS FOR TIME TO EVENT DATA

The time to first event will be summarised in terms of mean, standard deviation, median, minimum and maximum. The table of the estimated hazard rate will be presented, along with a Kaplan-Meier plot of the hazard function.

#### 9.1.3 ANALYSIS OF CONTINUOUS DATA

The absolute values and change from baseline in each endpoint will be summarised for each time point using N, mean, standard deviation, median, minimum and maximum.

#### 9.1.4 ANALYSIS FOR BINARY DATA

Binary data will be presented using counts and percentages. To calculate the percentage, the denominator will be the number of subjects with a non-missing value. These will be presented for each time point.

#### 9.1.5 ANALYSIS OF CATEGORICAL DATA

Categorical data will be summarized in terms of number and percentage of patients within each category at each visit. Shift tables of changes from baseline will also be presented.

#### 9.1.6 COMPARISON BETWEEN TREATMENTS

As there is only one cohort, those who are initiated on tofacitinib, there will be no formal comparison between treatment groups, although endpoints may be summarised by treatment subgroups (Section 6.6). All descriptive statistics will be presented overall and for all secondary analyses this will only be done using the data recorded when patients were taking tofacitinib.

#### 9.2 STATISTICAL ANALYSES

The statistical software SAS 9.3 (or higher) will be used to conduct the statistical analysis.

The results will be presented in tables and plots programmed within SAS.

Both the interim and final analyses will be performed using the methods described in this SAP. The outputs to be produced for the interim analysis will be flagged in the list of tables.

# 9.2.1 BACKGROUND AND DEMOGRAPHIC CHARACTERISTICS AND STUDY DISPOSITION

The Demographic and baseline variables will be summarised:

Continuous: Mean, standard deviation, median, minimum and maximum

Categorical: Frequency and Percentage of population.


This will include age, sex, height, weight, smoking history, smoking status, severity of disease, duration of disease, anti-citrullinated protein antibodies (ACPA) / RF, vaccination status, presence of Poor Prognostic Factors, comorbidities, co-medication and concomitant medication and will be based on the Full Analysis Set.

The number and percentage of patients at each time point will be provided along with reasons for withdrawal from the study. For patients who have discontinued to facitinib treatment but remain in the study, information on the treatments prescribed following study treatment (to facitinib) will be provided.

The baseline visit for each patient will be their Baseline (Enrollment) visit (Visit 1).

#### 9.2.2 PRIMARY ANALYSES

Each of the factors that will be included in the models for the primary analysis will be summarized by time point.

The Primary endpoint will be analysed as recurrent event data (as described in Section 9.1.1). The factors of interest as well as potential confounders (as described in Section 7.3.1 and section 6.3.3 respectively) will be included so as to determine whether they have an impact on the rate of treatment change. The population used for this analysis will be the FAS, including all visits (scheduled and unscheduled). The analysis will be repeated using the PPAS with visit windows as outlined in Section 12.1.1).

Escalations occurring in-between two planned visits will be assigned to visits using the visit windows provided in section 12.1.1. If two or more escalations fall into the same window, all escalations will be counted. Escalations, which are assigned to the baseline visit, will be counted under the Month 3 Visit, unless the escalation occurred before first tofacitinib treatment. Escalations, which fall outside the visit windows, will be assigned to the visit nearest to the Target Day. If two visits are equal distance from the escalation date in absolute value, the later visit should be used.

Sensitivity analyses, using both the FAS and PPAS, will be carried out with the covariates mentioned in section 7.3 along with the confounders mentioned above. An exploration of covariates will be carried out to assess any colinearity.

A further sensitivity analysis will be carried out using the FAS and PPAS population where treatment switches will be assigned to the visit prior to the date at which it occurred.


#### 9.2.3 SECONDARY ANALYSES

All secondary endpoints will be analysed using the SFAS.

Other subgroup analyses maybe carried out, these will be defined prior to database lock.

NOTE: Although a subject will be included in the analysis set regardless of their sequence of treatment, only data collected while a subject was on tofacitinib will be included in the secondary analyses. Methods used are described in Section 9.1.2 - 9.1.4.

#### 9.2.3.1 TIME TO FIRST TREATMENT ESCALATION

Time to first treatment escalation will be analysed as in Section 9.1.2 using the SFAS. Missing or incomplete dates will not be imputed (as per Section 8.1).

#### **9.2.3.2 RATE OF LDA**

Each definition of LDA (Section 7.1.2.2) will be presented as in Section 9.1.4, using the SFAS, only including data when patients were taking tofacitinib. Missing data will not be imputed (as per Section 8.2).

#### 9.2.3.3 RATE OF REMISSION

Each definition of Remission (Section 7.1.2.3) will be presented as in Section 9.1.4, using the SFAS, only including data when patients were taking to facitinib. Missing data will not be imputed (as per Section 8.2).

#### 9.2.3.4 CHANGE FROM BASELINE IN DAS28-4 (ESR) AND DAS28-4 (CRP)

Change from baseline in DAS28-4 (ESR) and DAS28-4 (CRP) will be presented and analysed as in Section 9.1.3, using the SFAS, only including data when patients were taking tofacitinib. Missing data will not be imputed (as per Section 8.2)

#### 9.2.3.5 CHANGE FROM BASELINE IN DURATION OF MORNING STIFFNESS

Duration of morning stiffness will be presented as in Section 9.1.3, using the SFAS, only including data when patients were taking tofacitinib. Missing data will not be imputed (as per Section 8.2)

#### 9.2.3.6 CHANGE FROM BASELINE IN FFBH

Change from baseline in FFbH score will be presented and analysed as in Section 9.1.3, using the SFAS, only including data when patients were taking tofacitinib. Missing data will not be imputed (as per Section 8.2)


#### 9.2.3.7 RATE OF FUNCTIONAL REMISSION

Rate of Functional Remission (Section 7.1.2.7) will be presented as in Section 9.1.4, using the SFAS, only including data when patients were taking to facitinib. Missing data will not be imputed (as per Section 8.2).

#### 9.2.3.8 CHANGE FROM BASELINE IN EQ-5D

Change from baseline in EQ-5D score (Section 7.1.2.8) will be presented and analysed as in Section 9.1.3, using the SFAS, only including data when patients were taking tofacitinib.

#### 9.2.3.9 CHANGE FROM BASELINE IN FACIT-FATIGUE

Change from baseline in FACIT-FATIGUE score (Section 7.1.2.9) will be presented and analysed as in Section 9.1.3, using the SFAS, only including data when patients were taking tofacitinib.

#### 9.2.3.10 DRUG SURVIVAL STATUS OF TOFACITINIB

Time to cease taking to facitinib (drug survival) will be analysed as per Section 9.1.2, using the SFAS. Missing data will not be imputed (as per Section 8.1).

#### 9.2.3.11 PATIENT'S SATISFACTION WITH DRUG TREATMENT

The Patient satisfaction is measured through a 5-point likert question asked at each visit and will be presented as in Section 9.1.5, using the FAS. At each visit, Visit X, only those who remained on tofacitinib at the previous visit, Visit X-1, will be presented. At each visit the satisfaction will be summarised split by those who remain on tofacitinib at Visit X and those who stop taking tofacitinib at Visit X.

#### 9.2.4 SAFETY ANALYSES

• Adverse events will be summarized according to Pfizer standards.

Two sets of 'All Causality' and 'Treatment Emergent' adverse events will be summarised:

The first set will contain adverse event data for subjects while they were taking tofacitinib either as a monotherapy or in combination with MTX (patients will be included in this group if they have taken MTX at any point in the study in combination tofacitinib regardless of duration). This AE table will summarise AEs under one treatment heading


for tofacitinib (which includes monotherapy and combination therapy with MTX). A drug lag of 28 days will be used to assign treatment emergence to tofacitinib. The second set will contain treatment emergent adverse events, which are related to tofacitinib and reported in a separate table.

Adverse events which occurred under another DMARD, following cessation of Tofacitinib, will only be listed and presented in a separate listing. AEs, which starts on the first day of a new treatment, e.g. Enbrel will be assigned to tofacitinib if the AE is within 28 days of tofacitinib. For non-Tofacitinib therapies a drug lag of 0 days will be applied. The AE will hence, also appear in the listing for other DMARDs as the AE started after the initiation of Enbrel. Therefore, any event which occurs during a 28 day lag of discontinuing tofacitinib will appear under tofacitinib in the tables and listings, and under the new treatment in the DMARD listing.

An all AE listing will show all AEs, individual rheumatologic therapies that are linked to the AE and whether the AE is tofacitinib treatment emergent.

#### **Treatment labels for reporting adverse events:**

Primary Adverse event table to assess AEs during to facitinib treatment:

tofacitinib

#### 9.2.5 SUBGROUP ANALYSIS

In addition to the analyses described above secondary endpoints will be analysed split by the subgroups described in section 6.6, as appropriate.

If additional subgroup analyses are needed, the details will be included as an amendment to this SAP prior to database release.

#### 9.2.6 SUMMARY OF ANALYSES

| Outcome | Analysis Set | Supports<br>Protocol<br>Objective<br>Number | Subgroups | Statistical<br>Method | Covariates/<br>Strata | Missing<br>Data |
|---|---|---|---|---|---|---|
| Number of<br>Treatment<br>Escalations | FAS | | | Cox-<br>Proportional<br>hazards with<br>recurrent events<br>(Section 9.1.1) | Covariates: DAS28-4(ESR) ≤ 3.2, ADAS28- 4(ESR) > 1.8, PtGA, PhyGA, | Imputation |


| | | | Pain, Satisfaction Confounders: Age, Gender, Duration of disease, Indicator of tofacitinib dose, Poor prognostic factors (PF) Indicator, Indicator of dose of MTX or combination partner, Indicator of dose of Glucocorticoids, Whether patient on 2nd or 3rd line treatment, Indicator of tolerability issues, Indicator of efficacy issues, comorbidities: Ischemic cardiovascular disease, Malignancies, Infections, Gastro disease, Osteoporosis, Depression (Note: will be assessed as individual covariates or as a composite, with 1 if a patient has any comorbidity or 0 otherwise, as appropriate). | |
|---|---|---|---|---|
| Number of<br>Treatment<br>Escalations | PPAS | Cox-<br>Proportional<br>hazards with<br>recurrent events<br>(Section 9.1.1) | Covariates: DAS28-4(ESR) ≤ 3.2, ΔDAS28- 4(ESR) > 1.8, PtGA, PhyGA, Pain, Satisfaction Confounders: Age, Gender, Duration of disease, Indicator of tofacitinib dose, Poor prognostic | No<br>Imputation |

| | | | | factors (PF) | |
|---|---|---|---|---|---|
| | | | | Indicator, | |
| | | | | Indicator of | |
| | | | | dose of MTX or combination | |
| | | | | partner, | |
| | | | | Indicator of | |
| | | | | dose of | |
| | | | | Glucocorticoids, | |
| | | | | Whether patient on 2 <sup>nd</sup> or 3 <sup>rd</sup> line | |
| | | | | treatment, | |
| | | | | Indicator of | |
| | | | | tolerability | |
| | | | | issues, | |
| | | | | Indicator of efficacy issues, | |
| | | | | comorbidities: | |
| | | | | Ischemic | |
| | | | | cardiovascular | |
| | | | | disease, | |
| | | | | Malignancies,<br>Infections, | |
| | | | | Gastro disease, | |
| | | | | Osteoporosis, | |
| | | | | Depression | |
| | | | | (Note: will be assessed as | |
| | | | | individual | |
| | | | | covariates or as | |
| | | | | a composite, | |
| | | | | with 1 if a | |
| | | | | patient has any comorbidity or | |
| | | | | 0 otherwise, as | |
| | | | | appropriate). | |
| Number of | FAS | | Cox- | Covariates: | No |
| Treatment | TAS | | Proportional | DAS28-4(ESR), | Imputation |
| Escalations | | | hazards with | ΔDAS28 | Imputation |
| (Sensitivity | | | recurrent events | 4(ESR), PtGA, | |
| Analysis) | | | (Section 9.1.1) | PhyGA, Pain, | |
| | | | , | Satisfaction,<br>Comorbidities | |
| | | | | (1 if patient has | |
| | | | | any | |
| | | | | comorbidity, 0 | |
| | | | | otherwise). | |
| | | | | Confounders: | |
| | | | | Age, Gender, | |
| | | | | Duration of | |
| | | | | disease, | |
| | | | | Indicator of tofacitinib dose, | |
| | | | | Poor prognostic | |
| | | | | factors (PF) | |
| | | | | Indicator, | |
| | | | | Indicator of | |
| | | | | dose of MTX or combination | |
| | | | | partner, | |
| | | i | | post orrest, | i l |


\_\_\_\_\_

| | | | Indicator of dose of Glucocorticoids, Whether patient on 2nd or 3rd line treatment, Indicator of tolerability issues, Indicator of efficacy issues, If the overall comorbidity covariate is significant the individual comorbidity covariates (Ischemic cardiovascular disease, Malignancies, Infections, Gastro disease, Osteoporosis, Depression) may be included as confounders instead as appropriate. | |
|---|---|---|---|---|
| Number of Treatment Escalations (Sensitivity Analysis) | PPAS | Cox-<br>Proportional<br>hazards with<br>recurrent events<br>(Section 9.1.1) | Covariates: DAS28-4(ESR), ADAS28- 4(ESR), PtGA, PhyGA, Pain, Satisfaction, Comorbidities (1 if patient has any comorbidity, 0 otherwise). Confounders: Age, Gender, Duration of disease, Indicator of tofacitinib dose, Poor prognostic factors (PF) Indicator, Indicator of dose of MTX or combination partner, Indicator of dose of Glucocorticoids, Whether patient on 2 <sup>nd</sup> or 3 <sup>rd</sup> line treatment, | No<br>Imputation |


| | | | Indicator of tolerability issues, Indicator of efficacy issues. If the overall comorbidity covariate is significant the individual comorbidity covariates (Ischemic cardiovascular disease, Malignancies, Infections, Gastro disease, Osteoporosis, Depression) may be included as confounders instead as appropriate. | |
|---|---|---|---|---|
| Number of Treatment Escalations (where treatment switch is assigned to prior visit – further sensitivity) | FAS | Cox-<br>Proportional<br>hazards with<br>recurrent events<br>(Section 9.1.1) | Covariates: DAS28-4(ESR) ≤ 3.2, ΔDAS28- 4(ESR) > 1.8, PtGA, PhyGA, Pain, Satisfaction Confounders: Age, Gender, Duration of disease, Indicator of tofacitinib dose, Poor prognostic factors (PF) Indicator, Indicator of dose of MTX or combination partner, Indicator of dose of Glucocorticoids, Whether patient on 2 <sup>nd</sup> or 3 <sup>rd</sup> line treatment, Indicator of tolerability issues, Indicator of efficacy issues, comorbidities: Ischemic cardiovascular disease, Malignancies, | Imputation |


| | | | Infections, Gastro disease, Osteoporosis, Depression (Note: will be assessed as individual covariates or as a composite, with 1 id a patient has any comorbidity or 0 otherwise, as appropriate). | |
|---|---|---|---|---|
| Number of Treatment Escalations (where treatment switch is assigned to prior visit further sensitivity) | PPAS | Cox-<br>Proportional<br>hazards with<br>recurrent events<br>(Section 9.1.1) | Covariates: DAS28-4(ESR) ≤ 3.2, ADAS28- 4(ESR) > 1.8, PtGA, PhyGA, Pain, Satisfaction Confounders: Age, Gender, Duration of disease, Indicator of tofacitinib dose, Poor prognostic factors (PF) Indicator, Indicator of dose of MTX or combination partner, Indicator of dose of Glucocorticoids, Whether patient on 2 <sup>nd</sup> or 3 <sup>rd</sup> line treatment, Indicator of tolerability issues, Indicator of efficacy issues, comorbidities: Ischemic cardiovascular disease, Malignancies, Infections, Gastro disease, Osteoporosis, Depression (Note: will be assessed as individual covariates or as a composite, with 1 id a patient has any | No<br>Imputation |


| | | | | comorbidity or 0 otherwise, as appropriate). | |
|---|---|---|---|---|---|
| Time to First<br>Treatment<br>Escalation | FAS | | Kaplan-Meier<br>Plots and Table<br>(Section 9.1.2) | | No<br>imputation |
| Rate of LDA | FAS, including only data collected with patient remained on tofacitinib | Therapy Sequence, RA Medication History, Switch Status, Number of Treatment Switches (Section 6.6) | Summary<br>Tables (Section<br>9.1.4) | | No<br>imputation |
| Rate of<br>Remission | FAS, including only data collected with patient remained on tofacitinib | Therapy Sequence, RA Medication History, Switch Status, Number of Treatment Switches (Section 6.6) | Summary<br>Tables (Section<br>9.1.4) | | No<br>imputation |
| Change from baseline DAS28-4 | FAS, including only data collected with patient remained on tofacitinib | Therapy Sequence, RA Medication History, Switch Status, Number of Treatment Switches (Section 6.6) | Summary<br>Tables (Section<br>9.1.3) | | No<br>imputation |
| Change from baseline in Morning Stiffness | FAS, including only data collected with patient remained on tofacitinib | Therapy Sequence, RA Medication History, Switch Status, Number of Treatment Switches (Section 6.6) | Summary<br>Tables (Section<br>9.1.3) | | No<br>imputation |
| Change from baseline in | FAS, including only data | Therapy<br>Sequence, | Summary<br>Tables (Section | | No<br>imputation |
| FFbH<br>Final Version | collected with | RA 07-AUG-2023 | 9.1.3) | _ | e 41 of 48 |


| | patient | Medication | | | |
|---|---|---|---|---|---|
| | remained on | History, | | | |
| | tofacitinib | Switch | | | |
| | | Status, | | | |
| | | Number of | | | |
| | | Treatment | | | |
| | | Switches | | | |
| | | (Section 6.6) | | | |
| Rate of | FAS, including | Therapy | Summary | | No |
| functional | only data | Sequence, | Tables (Section | | imputation |
| remission in | collected with | RA | 9.1.4) | | 1 |
| FFbH | patient | Medication | , | | |
| | remained on | History, | | | |
| | tofacitinib | Switch | | | |
| | | Status, | | | |
| | | Number of | | | |
| | | Treatment | | | |
| | | Switches | | | |
| | | (Section | | | |
| | T. C. 1 11 | 6.6) | ~ | | 2.7 |
| Change from | FAS, including | Therapy | Summary | | No |
| baseline in EQ-<br>5D score | only data collected with | Sequence,<br>RA | Tables (Section | | imputation |
| 3D score | patient | Medication | 9.1.3) | | |
| | remained on | History, | | | |
| | tofacitinib | Switch | | | |
| | toracitino | Status, | | | |
| | | Number of | | | |
| | | Treatment | | | |
| | | Switches | | | |
| | | (Section | | | |
| | | 6.6) | | | |
| Change from | FAS, including | Therapy | Summary | | No |
| baseline in | only data | Sequence, | Tables (Section | | imputation |
| FACIT score. | collected with | RA | 9.1.3) | | |
| | patient | Medication | | | |
| | remained on | History, | | | |
| | tofacitinib | Switch | | | |
| | | Status,<br>Number of | | | |
| | | Treatment | | | |
| | | Switches | | | |
| | | (Section | | | |
| | | 6.6) | | | |
| Drug Survival | FAS | , | Kaplan-Meier | | No |
| | | | Plots and Table | | imputation |
| | | <br> | (Section 9.1.2) | | _ |
| Patient's | FAS, | Therapy | Summary | - | No |
| Satisfaction | | Sequence, | Tables (Section | | imputation |
| with Drug | | RA | 9.1.5) | | |
| Treatment | | Medication | | | |
| | | History, | | | |
| | | Switch | | | |
| | | Status, | | | |
| | | Number of Treatment | | | |
| | | Switches | | | |
| | | Switches | | | |


| (Section |
|----------|
| 6.6) |

# 10 LIST OF TABLES AND TABLE SHELLS

To be presented in a separate document.

#### 11 REFERENCES

- 1 Strand V, Singh JA. Improved health-related quality of life with effective disease modifying antirheumatic drugs: evidence from randomized controlled trials. The American journal of managed care. 2007;13 Suppl 9:S237-51. Epub 2007/01/12.
- 2 Gullick NJ, Scott DL. Co-morbidities in established rheumatoid arthritis. Best Pract Res Clin Rheumatol. 2011 Aug;25 (4):469-83
- 3 Brown K. Rheumatoid Lung Disease. Proc Am Thorac Soc 2007;4:443–448
- 4 Gerhold K, Richter A, Schneider M, Bergerhausen H-J et al. Health-related quality of life in patients with long-standing rheumatoid arthritis in the era of biologics: data from the German biologics register RABBIT Rheumatology (Oxford) 2015;54(10):1858–1866
- 5 Boonen A, Severens JL. The burden of illness of rheumatoid arthritis. Clin Rheumatol. 2011;30 Suppl 1:S3–8
- 6 Zhang W, Anis AH. The economic burden of rheumatoid arthritis: beyond health care costs. Clin Rheumatol. 2011;30 Suppl 1:S25–32. CT24-GSOP-RF03 NI Study Protocol Template; Version 3.0, Effective Date 10-Oct-2014 Pfizer Confidential Page 47 of 50 Tofacitinib citrate A3921302 OBSERVATIONAL PLAN NON-INTERVENTIONAL STUDY Final, 27 June 2017
- 7 Emery P. Evidence supporting the benefit of early intervention in rheumatoid arthritis. J Rheumatol Suppl. 2002 Nov;66:3-8.
- 8 Pincus T. Rheumatoid arthritis: a medical emergency? Scand J Rheumatol Suppl. 1994;100:21-30.
- 9 Nell VP, Machold KP, Eberl G, et al. Benefit of very early referral and very early therapy with disease modifying anti-rheumatic drugs in patients with early rheumatoid arthritis. Rheumatology (Oxford) 2004;43:906–14.
- 10 van Nies JA, Krabben A, Schoones JW, et al. What is the evidence for the presence of a therapeutic window of opportunity in rheumatoid arthritis? A systematic literature review. Ann Rheum Dis 2014 May;73(5):861-70.
- 11 Grigor C, Capell H, Stirling A, et al. Effect of a treatment strategy of tight control for rheumatoid arthritis (the TICORA study): a singleblind randomized controlled trial. Lancet 2004;364:263–9.
- 12 Smolen, J. S., R. Landewe, J. Bijlsma, G. Burmester, K. Chatzidionysiou, M. Dougados, J. Nam, *et al.* "Eular Recommendations for the Management of Rheumatoid Arthritis with Synthetic and


Biological Disease-Modifying Antirheumatic Drugs: 2016 Update." [In eng]. *Ann Rheum Dis* 76, no. 6 (Jun 2017): 960-77

- 13 Felson DT, Smolen JS, Wells G, et al. American college of rheumatology/European league against rheumatism provisional definition of remission in rheumatoid arthritis for clinical trials. Ann Rheum Dis 2011;70:404–13.
- 14 Albrecht et al. 2016 Klinische Remission bei rheumatoider Arthritis Daten aus der Früharthritiskohortenstudie CAPEA Z. Rheumatol 75:90-96).
- 15 Albrecht et al. 2017, Versorgung der rheumatoiden Arthritis 2014 Aktuelle Daten aus der Kerndokumentation, Z. Rheumatol 76:50-57
- 16 Louder MA, Singh A, Saverno K, Cappelleri JC, Aten AJ et al. Patient Preferences Regarding Rheumatoid Arthritis Therapies: A Conjoint Analysis. Am Health Drug Benefits. 2016;9(2):84-93
- 17 Krüger K, Alten R, Schiffner-Rohe J, Behmer OS, Schiffhorst G, J. Rellecke J, Nolting H. D. Patient preference in the choice of disease modifying anti-rheumatic drugs. Poster presented at the EULAR Annual European Congress of Rheumatology, Rome, Italy, June 10-13, 2015
- 18 A3921302\_ObservationalPlan\_Finalv1.1\_23Aug2017.docx


### 12 APPENDICES

# 12.1 APPENDIX 1: DATA DERIVATION DETAILS

# 12.1.1 A1.1 DEFINITION AND USE OF VISIT WINDOWS IN REPORTING

Visit windows will be used for efficacy variables, and for any safety displays that display by month. The visit windows for the analysis defined in the table differ from that outlined in the protocol. The analysis visit windows will be M1, M3 $\pm$ 14 days, all subsequent visits MX  $\pm$  28 days.

| Table 11.1: Visit windows | | |
|---------------------------|------------|-------------------------|
| Visit Label | Target Day | Definition [Day window] |
| Enrolment | 1 | 1 |
| Month 3 | 91 | 77 to 105 |
| Month 6 | 182 | 154 to 210 |
| Month 9 | 273 | 245 to 301 |
| Month 12 | 365 | 337 to 393 |
| Month15 | 456 | 428 to 484 |
| Month18 | 547 | 519 to 575 |
| Month 21 | 638 | 610 to 666 |
| Month 24 | 730 | 702 to 758 |

For the lab values, if the calculated study day for the labelled baseline visit is not study Day 1, but falls within 40 days before the start of the study dosing, then that data should be used for the baseline instead of leaving baseline missing.

For the other values, if the calculated study day for the labelled baseline visit is not study Day 1, but falls before the start of the study dosing, then that data should be used for the baseline instead of leaving baseline missing.

If baseline is missing there will be no imputation and although the subject's data will be included in summary data it will not be included in any change from baseline analyses.

If two or more visits fall into the same window, keep the one closest to the Target Day. If two visits are equal distance from the Target Day in absolute value, the later visit should be used.

For the primary endpoint analysis, escalations occurring in-between two planned visits will be assigned to visits using the visit windows described above. If two or more escalations


fall into the same window, all escalations will be counted. Escalations, which are assigned to the baseline visit, will be counted under the Month 3 Visit, unless the escalation occurred before first tofacitinib treatment. Escalations, which fall outside the visit windows, will be assigned to the visit nearest to the Target Day. If two visits are equal distance from the escalation date in absolute value, the later visit should be used.

(Safety analysis may follow Pfizer standard)

# 12.1.2 DEFINITION OF TREATMENT ESCALATIONS

Table 11.2 provides an overview of all possible treatment switch combinations relevant for the analysis of the primary endpoint and defines the type of escalations, e.g., whether the treatment switch relates to a step-up, step-down or termination.


Table 12.2: Definition of treatment escalations Therapy\*> Mono Mono tsDMARD MonoTNFi ComboTNFi Therapy Mono Mono bDMARD Combo+ Combo tsDMARD Combo Tofa csDMARD csDMARD +csDMARD +csDMARD bDMARD+ Stop csDMARD Step-up MonoTofa Step-up Step-down Step-up Step-up Step-up Step-up Step-up Treatment termination Step-up if different Mono Step-up Step-down Step-up Step-up Step-up Step-up Step-up Step-up Treatment tsDMARD tsDMARD termination Mono Step-up Step-up Step-up Step-up if Step-up Step-up Step-up Step-up Step-up Treatment different csDMARD termination csDMARD Step-up Step-up Step-down Step-up if Step-up Step-up MonoTNFi Step-up Step-up Step-up Treatment termination different TNFi Mono Step-up Step-up Step-down Step-up Step-up if different Step-up Step-up Step-up Step-up Treatment **bDMARD bDMARD** termination Combo+ Step-Step-up Step-down Step-up Step-up Step-up if Step-up Step-up Step-up Treatment **csDMARD** different down termination csDMARD Step-up if different Step-down Step-up Step-up if different Combo Step-up Step-up Step-up Step-up Step-up Treatment tsDMARD tsDMARD: tsDMARD or termination +csDMARD Step-down otherwise csDMARD Step-up Step-up Step-down, if Step-down Step-up Step-up Step-up Step-up if Step-up if Combo Treatment TNFi+ same TNFi. different different termination csDMARD Step-up if csDMARD/TN bDMARD or different TNFi csDMARD Step up Step down if same Step up Step up Combo Step up Step down Step up Step up Step up if Treatment bDMARD+ bDMARD; Step-up different termination csDMARD bDMARD or otherwise csDMARD \*) Definitions: Mono tsDMARD= Monotherapy any tsDMARD other than Tofa Combo tsDMARD + csDMARD= Combination therapy tsDMARD

\*) Definitions:

Mono tsDMARD= Monotherapy any tsDMARD other than Tofa
Mono csDMARD= Monotherapy any csDMARD

Combo= Combination

Mono TNFi= Monotherapy any TNFi

Tofa= tofacitinib

Mono bDMARD= Monotherapy any bDMARD other than TNFi

TNFi= Tumor Necrosis Factor Inhibitor

Mono Tofa= Combination therapy tofacitinib with any csDMARD

Mono Tofa= Monotherapy tofacitinib

Combo csDMARD= Combination therapy tofacitinib + any csDMARD

Combo tsDMARD + csDMARD= Combination therapy tsDMARD other than tofacitinib + any csDMARD

Combo TNFi + csDMARD= Combination therapy any TNFi+ any csDMARD

Combo bDMARD + csDMARD= Combination therapy bDMARD other than TNFi+ anycsDMARD


**DocuSign** 

# PDD

# PD

# PPD

## LEGAL DISCLOSURE

By electronically signing a document provided by AMS through the Docusign electronic signatures system, I expressly consent to the use of the system and confirm that I understand my signature will have the same binding effect as a handwritten signature.

I also confirm that the email address I am using is a valid and personalized email address, appropriate for identification and notification of myself as a Signee of a document. I will inform AMS in the case that my email address changes.

# ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, AMS Advanced Medical Services GmbH (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

# Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

# Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

# Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

# All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

### **How to contact AMS Advanced Medical Services GmbH:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: docusign@ams-europe.com

# To advise AMS Advanced Medical Services GmbH of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at docusign@ams-europe.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

# To request paper copies from AMS Advanced Medical Services GmbH

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to docusign@ams-europe.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

# To withdraw your consent with AMS Advanced Medical Services GmbH

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to docusign@ams-europe.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

# Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

# Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and

• Until or unless you notify AMS Advanced Medical Services GmbH as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by AMS Advanced Medical Services GmbH during the course of your relationship with AMS Advanced Medical Services GmbH.